CLINICAL TRIAL: NCT03984201
Title: Accelerated Theta Burst in Chronic Pain: A Biomarker Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The site was unable to recruit participants.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Nolan R, Assistant Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 48366
Record Dates: First submitted 2019-05-30; First posted 2019-06-12 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Repetitive Transcranial Magnetic Stimulation (rTMS); Accelerated Theta Burst Stimulation (aTBS); Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT)
MeSH Terms: conditions — Chronic Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Blinded, randomized control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- iTBS over L-DLPFC to dACC (Active Comparator): Participants will receive iTBS (intermittent theta burst stimulation) to the left dorsal lateral prefrontal cortex (L-DLPFC) with high connectivity to the dorsal anterior cingulate cortex (dACC). The L-DLPFC will be targeted utilizing the Localite neuronavigation system. Stimulation intensity will be standardized at 90% of resting motor threshold adjust to the skull to cortical surface distance.
  Stimulation will be delivered to L-DLPFC using the MagPRo stimulator.
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS)
- iTBS over L-DLPFC to sgACC (Active Comparator): Participants will receive iTBS (intermittent theta burst stimulation) to the left dorsal lateral prefrontal cortex (L-DLPFC) with high connectivity to the subgenual cingulate cortex (sgACC). The L-DLPFC will be targeted utilizing the Localite neuronavigation system. Stimulation intensity will be standardized at 90% of resting motor threshold adjust to the skull to cortical surface distance.
  Stimulation will be delivered to L-DLPFC using the MagPRo stimulator.
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS)
- Sham iTBS over L-DLPFC (Sham Comparator): Participants will receive sham iTBS (intermittent theta burst stimulation) to the left DLPFC. The L-DLPFC will be targeted utilizing the Localite neuronavigation system.
  Sham stimulation will be delivered to L-DLPFC using the MagPRo stimulator.
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS)

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation (iTBS) — Participants will receive active or sham transcranial magnetic stimulation delivered to the L-DLPFC.
  Other Names: Accelerated Theta Burst Stimulation (aTBS); Repetitive Transcranial Magnetic Stimulation (rTMS)

SUMMARY:
This study evaluates an accelerated schedule of theta-burst stimulation using a transcranial magnetic stimulation device for chronic pain. In this double blind, randomized control study, participants will be randomized to the treatment group to receive accelerated theta-burst stimulation or to a control group. All participants will be offered the open-label, active treatment 4 week prior to completing the initial 5 days of treatment.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an established technology as therapy for treatment-resistant depression and has been utilized to treat persons suffering from chronic pain. The approved method for treatment is 10Hz stimulation for 40 min over the left dorsolateral prefrontal cortex (L-DLPFC). This methodology has been very successful in real world situations. The limitations of this approach include the duration of the treatment (approximately 40 minutes per treatment session). Recently, researchers have aggressively pursued modifying the treatment parameters to reduce treatment times with some preliminary success. This study intends to further modify the parameters to create a more rapid form of the treatment and look at the change in neuroimaging biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients need to meet at least a 4/10 on a clinical pain rating scale and/or fulfill fibromyalgia diagnostic criteria on the 2010 Fibromyalgia Diagnostic Criteria (Wolfe et al., 2010)
2. Age 18 - 70
3. Right-handed
4. Agree to having fMRI scans as well as rTMS sessions
5. Proficiency in English sufficient to complete questionnaires / follow instructions during fMRI assessments and treatment
6. Women of childbearing potential must agree to use adequate contraception prior to study entry and continue this for the duration of the study
7. Participants may continue antidepressant regimen, but must be stable for 6 weeks prior to enrollment in the study. Antidepressant must be of the SSRI class only (if currently on a different antidepressant, patients will be switched to an SSRI). They must maintain that same antidepressant regimen throughout the study duration.

Exclusion Criteria:

1. History of MI, CABG, CHF, or other cardiac history.
2. Any condition that would contraindicate MRI (such as ferromagnetic metal in the body)
3. Pregnancy or breastfeeding
4. Any neurological condition, history of epilepsy, history of rTMS failure with FDA approved rTMS parameters, history of any implanted device or psychosurgery for depression, history of receiving ECT. OCD, narcolepsy or any additional significant neurological disorder as determined by the PI.
5. Autism spectrum disorder
6. Inability to stop taking medication contraindicated with treatment
7. Any significant psychiatric disorder as identified on the Mini International Neuropsychiatric Interview and determined by the PI
8. A positive urine toxicology screen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in the Brief Pain Inventory (BPI) score | Pre-treatment, immediately post-treatment
  A self-report measure designed to enable investigators to easily obtain sensitive measures of the degree of depression and individual is experiencing.
  Scoring:
  1. Pain Severity Score: This is calculated by adding the scores for questions 2, 3, 4 and 5 and then dividing by 4. This gives a severity score out of 10.
  2. Pain Interference Score: This is calculated by adding the scores for questions 8a, b, c, d, e, f and g and then dividing by 7. This gives an interference score out of 10.
Change in the McGill Pain Questionnaire score | Pre-treatment, immediately post-treatment
  A self-report questionnaire that allows individuals that assesses the quality and intensity of pain that is experienced. The pain rating index has 2 subscales: sensory subscale with 11 words, and affective subscale with 4 words. These items are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate and 3 = severe. There's also one item for present pain intensity and one item for a 10cm visual analogue scale for average pain.

SECONDARY OUTCOMES:
Change in the Montgomery Asberg Depression Rating Scale (MADRS) score | Pre-treatment, immediately post-treatment, 2 weeks post-treatment, 4 weeks post-treatment
  A ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders.
  Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60; 0 to 6 - normal, symptom absent; 7 to 19 - mild depression; 20 to 34 - moderate depression; >34 - severe depression.
Change in teh Hamilton Rating Scale for Depression (HAM-17) score | Pre-treatment, immediately post-treatment, 2 weeks post-treatment, 4 weeks post-treatment
  A provider administered questionnaire used to assess remission and recovery from depression. in general the higher the total score the more severe the depression. HAM-D score level of depression: 10-13 mild; 14-17 mild to moderate; >17 moderate to severe.
Change in the Pain Catastrophizing Scale (PCS) score | Pre-treatment, immediately post-treatment, 2 weeks post-treatment, 4 weeks post-treatment
  A self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52 that measures a person's catastrophizing of pain. A higher score indicates a higher level of pain catastrophizing.
Change in functional connectivity as measured by Functional Magnetic Resonance Imaging (fMRI) | Pre-treatment, immediately post-treatment, 4 weeks post-treatment
  Participants will have fMRI scans both before the first treatment (baseline) and after the aiTBS course. The MRI scans will be used to identify potential biomarkers for antidepressant response and pain response, as well as identify aiTBS-induced changes in functional connectivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avery DH, Zarkowski P, Krashin D, Rho WK, Wajdik C, Joesch JM, Haynor DR, Buchwald D, Roy-Byrne P. Transcranial magnetic stimulation in the treatment of chronic widespread pain: a randomized controlled study. J ECT. 2015 Mar;31(1):57-66. doi: 10.1097/YCT.0000000000000125. PMID 24755729
- [Background] Baeken C, Marinazzo D, Everaert H, Wu GR, Van Hove C, Audenaert K, Goethals I, De Vos F, Peremans K, De Raedt R. The Impact of Accelerated HF-rTMS on the Subgenual Anterior Cingulate Cortex in Refractory Unipolar Major Depression: Insights From 18FDG PET Brain Imaging. Brain Stimul. 2015 Jul-Aug;8(4):808-15. doi: 10.1016/j.brs.2015.01.415. Epub 2015 Feb 7. PMID 25744500
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Bonelli RM, Cummings JL. Frontal-subcortical circuitry and behavior. Dialogues Clin Neurosci. 2007;9(2):141-51. doi: 10.31887/DCNS.2007.9.2/rbonelli. PMID 17726913
- [Background] Borckardt JJ, Nahas Z, Koola J, George MS. Estimating resting motor thresholds in transcranial magnetic stimulation research and practice: a computer simulation evaluation of best methods. J ECT. 2006 Sep;22(3):169-75. doi: 10.1097/01.yct.0000235923.52741.72. PMID 16957531
- [Background] Cieslik EC, Zilles K, Caspers S, Roski C, Kellermann TS, Jakobs O, Langner R, Laird AR, Fox PT, Eickhoff SB. Is there "one" DLPFC in cognitive action control? Evidence for heterogeneity from co-activation-based parcellation. Cereb Cortex. 2013 Nov;23(11):2677-89. doi: 10.1093/cercor/bhs256. Epub 2012 Aug 23. PMID 22918987
- [Background] Connolly KR, Helmer A, Cristancho MA, Cristancho P, O'Reardon JP. Effectiveness of transcranial magnetic stimulation in clinical practice post-FDA approval in the United States: results observed with the first 100 consecutive cases of depression at an academic medical center. J Clin Psychiatry. 2012 Apr;73(4):e567-73. doi: 10.4088/JCP.11m07413. PMID 22579164
- [Background] Duprat R, Desmyter S, Rudi de R, van Heeringen K, Van den Abbeele D, Tandt H, Bakic J, Pourtois G, Dedoncker J, Vervaet M, Van Autreve S, Lemmens GM, Baeken C. Accelerated intermittent theta burst stimulation treatment in medication-resistant major depression: A fast road to remission? J Affect Disord. 2016 Aug;200:6-14. doi: 10.1016/j.jad.2016.04.015. Epub 2016 Apr 19. PMID 27107779
- [Background] Gamboa OL, Antal A, Moliadze V, Paulus W. Simply longer is not better: reversal of theta burst after-effect with prolonged stimulation. Exp Brain Res. 2010 Jul;204(2):181-7. doi: 10.1007/s00221-010-2293-4. Epub 2010 Jun 22. PMID 20567808
- [Background] George MS, Ketter TA, Parekh PI, Rosinsky N, Ring H, Casey BJ, Trimble MR, Horwitz B, Herscovitch P, Post RM. Regional brain activity when selecting a response despite interference: An H2 (15) O PET study of the stroop and an emotional stroop. Hum Brain Mapp. 1994;1(3):194-209. doi: 10.1002/hbm.460010305. PMID 24578040
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Taylor JJ, Short EB. The expanding evidence base for rTMS treatment of depression. Curr Opin Psychiatry. 2013 Jan;26(1):13-8. doi: 10.1097/YCO.0b013e32835ab46d. PMID 23154644
- [Background] Grimm S, Beck J, Schuepbach D, Hell D, Boesiger P, Bermpohl F, Niehaus L, Boeker H, Northoff G. Imbalance between left and right dorsolateral prefrontal cortex in major depression is linked to negative emotional judgment: an fMRI study in severe major depressive disorder. Biol Psychiatry. 2008 Feb 15;63(4):369-76. doi: 10.1016/j.biopsych.2007.05.033. Epub 2007 Sep 21. PMID 17888408
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Kreuzer PM, Schecklmann M, Lehner A, Wetter TC, Poeppl TB, Rupprecht R, de Ridder D, Landgrebe M, Langguth B. The ACDC pilot trial: targeting the anterior cingulate by double cone coil rTMS for the treatment of depression. Brain Stimul. 2015 Mar-Apr;8(2):240-6. doi: 10.1016/j.brs.2014.11.014. Epub 2014 Nov 29. PMID 25541389
- [Background] Lan MJ, Chhetry BT, Liston C, Mann JJ, Dubin M. Transcranial Magnetic Stimulation of Left Dorsolateral Prefrontal Cortex Induces Brain Morphological Changes in Regions Associated with a Treatment Resistant Major Depressive Episode: An Exploratory Analysis. Brain Stimul. 2016 Jul-Aug;9(4):577-83. doi: 10.1016/j.brs.2016.02.011. Epub 2016 Mar 2. PMID 27017072
- [Background] Larson J, Munkacsy E. Theta-burst LTP. Brain Res. 2015 Sep 24;1621:38-50. doi: 10.1016/j.brainres.2014.10.034. Epub 2014 Oct 27. PMID 25452022
- [Background] Lee SJ, Kim DY, Chun MH, Kim YG. The effect of repetitive transcranial magnetic stimulation on fibromyalgia: a randomized sham-controlled trial with 1-mo follow-up. Am J Phys Med Rehabil. 2012 Dec;91(12):1077-85. doi: 10.1097/PHM.0b013e3182745a04. PMID 23159954
- [Background] Lefaucheur JP. The use of repetitive transcranial magnetic stimulation (rTMS) in chronic neuropathic pain. Neurophysiol Clin. 2006 May-Jun;36(3):117-24. doi: 10.1016/j.neucli.2006.08.002. Epub 2006 Aug 23. PMID 17046606
- [Background] Li CT, Chen MH, Juan CH, Huang HH, Chen LF, Hsieh JC, Tu PC, Bai YM, Tsai SJ, Lee YC, Su TP. Efficacy of prefrontal theta-burst stimulation in refractory depression: a randomized sham-controlled study. Brain. 2014 Jul;137(Pt 7):2088-98. doi: 10.1093/brain/awu109. Epub 2014 May 10. PMID 24817188
- [Background] Oberman L, Edwards D, Eldaief M, Pascual-Leone A. Safety of theta burst transcranial magnetic stimulation: a systematic review of the literature. J Clin Neurophysiol. 2011 Feb;28(1):67-74. doi: 10.1097/WNP.0b013e318205135f. PMID 21221011
- [Background] Ochsner, K. N., & Gross, J. J. (2005). Putting the ' I ' and the ' Me ' in emotion regulation : Reply to Northoff, (xx), 6613. https://doi.org/10.1016/j.tics.2005.06.005
- [Background] Ohayon MM. Specific characteristics of the pain/depression association in the general population. J Clin Psychiatry. 2004;65 Suppl 12:5-9. PMID 15315471
- [Background] Onghena P, Van Houdenhove B. Antidepressant-induced analgesia in chronic non-malignant pain: a meta-analysis of 39 placebo-controlled studies. Pain. 1992 May;49(2):205-219. doi: 10.1016/0304-3959(92)90144-Z. PMID 1535121
- [Background] Smolen P, Zhang Y, Byrne JH. The right time to learn: mechanisms and optimization of spaced learning. Nat Rev Neurosci. 2016 Feb;17(2):77-88. doi: 10.1038/nrn.2015.18. PMID 26806627
- [Background] Taylor JJ, Borckardt JJ, Canterberry M, Li X, Hanlon CA, Brown TR, George MS. Naloxone-reversible modulation of pain circuitry by left prefrontal rTMS. Neuropsychopharmacology. 2013 Jun;38(7):1189-97. doi: 10.1038/npp.2013.13. Epub 2013 Jan 11. PMID 23314221
- [Background] Taylor JJ, Borckardt JJ, George MS. Endogenous opioids mediate left dorsolateral prefrontal cortex rTMS-induced analgesia. Pain. 2012 Jun;153(6):1219-1225. doi: 10.1016/j.pain.2012.02.030. Epub 2012 Mar 22. PMID 22444187
- [Background] Tendler A, Roth Y, Barnea-Ygael N, Zangen A. How to Use the H1 Deep Transcranial Magnetic Stimulation Coil for Conditions Other than Depression. J Vis Exp. 2017 Jan 23;(119):55100. doi: 10.3791/55100. PMID 28190035
- [Background] Vanneste S, Ost J, Langguth B, De Ridder D. TMS by double-cone coil prefrontal stimulation for medication resistant chronic depression: a case report. Neurocase. 2014;20(1):61-8. doi: 10.1080/13554794.2012.732086. Epub 2012 Oct 11. PMID 23058173
- [Background] Williams NR, Sudheimer KD, Bentzley BS, Pannu J, Stimpson KH, Duvio D, Cherian K, Hawkins J, Scherrer KH, Vyssoki B, DeSouza D, Raj KS, Keller J, Schatzberg AF. High-dose spaced theta-burst TMS as a rapid-acting antidepressant in highly refractory depression. Brain. 2018 Mar 1;141(3):e18. doi: 10.1093/brain/awx379. No abstract available. PMID 29415152
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783